CLINICAL TRIAL: NCT05950243
Title: COVID-19 Disease & Vaccine Survey in Sub-Saharan Africa
Brief Title: COVID-19 Disease & Vaccine Survey in Africa
Status: Completed | Type: Observational
Sponsor: Salem Anaesthesia Pain Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: SalemAnes2021 COVID Africa
Record Dates: First submitted 2023-07-16; First posted 2023-07-18 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: COVID-19; Vaccine Hesitancy
Keywords: COVID-19
MeSH Terms: conditions — COVID-19; Vaccination Hesitancy | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Urban population Africa: Urban population in sub-Saharan Africa
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaire survey for data collection

SUMMARY:
The COVID-19 pandemic is a public health concern; for which the WHO recommends protective measures and vaccination. There is inadequate data on the impact of COVID-19 vaccination and control measures in Africa. This survey is collecting data about people's knowledge, attitude and compliance regarding COVID-19 disease and vaccines.

DETAILED DESCRIPTION:
The coronavirus disease 2019 (COVID-19) pandemic remains a major public health concern. There is inadequate data on the epidemiology of COVID-19 in Africa. There are emerging COVID-19 variants with high transmissibility and morbidity. The World Health Organization (WHO) recommends protective measures and vaccination; for the control of COVID-19. There is inadequate data on the impact of COVID-19 vaccination and control measures in many nations in Africa.

This study is a survey of specific urban populations in sub-Saharan Africa. The anonymized survey is collecting data about people's knowledge and attitude regarding COVID-19 disease or control measures. The survey is also collecting data about people's knowledge, attitude and compliance regarding COVID-19 vaccines. The study uses a validated questionnaire to collect data. The study aims to inform and improve COVID-19 management or control in Africa.

ELIGIBILITY:
Inclusion Criteria:

* urban population in Africa
* people in sub-Saharan Africa town

Exclusion Criteria:

* rural population
* people outside sub-Saharan Africa

Ages: 9 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Urban population in selected sub-Saharan African town or city
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2021-01-02 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Percentage of people who know about COVID-19 prevention | 6 months
  Percentage of people who know about COVID-19 preventive measures
Percentage of people who received COVID-19 vaccination | 6 months
  Percentage of people who received COVID-19 vaccination, 1st and 2nd doses

CONTACTS AND LOCATIONS:
Overall Officials: Olu Bamgbade, MD,FRCPC, Principal Investigator — Salem Anaesthesia Pain Clinic
Locations (1):
- Salem Anaesthesia Pain Clinic, Surrey, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No